CLINICAL TRIAL: NCT00351403
Title: Individually Adapted Therapy Duration From 24 to 72 Weeks for the Treatment of a Chronic Hepatitis C Genotype 1 Infection With Peginterferon Alfa-2b Plus Ribavirin in Dependence of the Initial Concentration and the Decline of the HCV RNA
Brief Title: Individually Adapted Therapy Duration for the Treatment of Chronic Hepatitis C Genotype 1 Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: FGK Clinical Research GmbH (Industry)
Collaborators: University Hospital, Saarland (Other)
Responsible Party: Christoph Sarrazin, MD, PhD, Universitätsklinikum des Saarlandes
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INDIV-2; 2006-000358-38 (EudraCT Number)
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2010-02

CONDITIONS: Hepatitis C, Chronic
Keywords: Chronic HCV infection; Genotype 1; Individually adapted therapy; Peginterferon alfa-2b; Ribavirin; Sustained viral response (SVR)
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individualized therapy (Experimental): Lengh of therapy depends on time point when no HCV RNA is detectable in blood with Versant HCV Qualitative assay.
  Interventions: Drug: Ribavirin; Drug: Peginterferon alfa 2b
- Historical control (Other): 48 week standard therapy
  Interventions: Drug: Ribavirin; Drug: Peginterferon alfa 2b

INTERVENTIONS:
Drug: Ribavirin — Rebetol 200 mg: applied as hard capsule
Drug: Peginterferon alfa 2b — PegIntron (50/80/100/120/150 microgram): applied by injection

SUMMARY:
Patients with chronic hepatitis C genotype 1 virus infection are usually treated with Interferon alfa plus Ribavirin over 48 weeks. For some patients this might be too long, for others too short. An individually adapted therapy length from 24 to 72 weeks will be determined in dependence of the initial virus load and the time to HCV RNA negativity.

The primary objective is to compare the cumulative rate of the sustained viral response (SVR) of the patients with the individually adapted therapy duration to the SVR rates of a historic patient collective under the 48 week standard therapy.

DETAILED DESCRIPTION:
Further objectives of this trial are:

To record the tolerance of the therapy with Peginterferon alfa-2b plus Ribavirin over 72 weeks inclusive the adverse reactions and the withdrawal rates.

To evaluate the biochemical response to the treatment (ALT values during and after the therapy) in comparison to the virological response to the treatment.

To evaluate the validity of the withdrawal rules of this trial at week 12 and 24 in comparison to the 2-log-rule and a qualitative detection of the HCV RNA at week 24 with a detection limit of 50 IU/ml.

To evaluate the impact of the HCV RNA concentration before the therapy, and the HCV kinetic during the therapy on the response to the treatment in the different groups.

To evaluate the impact of the serum concentration of Ribavirin on anaemia and the virological therapy response, as well as the dependence of the serum concentration of Ribavirin on the creatinine clearance in comparison to the body weight.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a chronic HCV infection (HCV antibodies and HCV RNA positive)
* Presence of a HCV genotype 1 infection
* Presence of a compensated liver disease satisfying following hematological and biochemical minimum criteria: - Hemoglobin value >= 13 g/dl in men, >= 12 g/dl in women - Leukocytes >= 3.000/mm3 or neutrophile granulocytes > 1.500/mm3 - Thrombocytes > 80.000/mm3
* Total bilirubin in the normal range
* Albumin in the normal range
* Serum creatinine in the normal range THS in the normal range
* Exclusion of an autoimmune hepatitis
* Alpha-Fetoprotein in the normal range
* Negative HIV test
* Negativity of Hepatitis B surface antigens (Hbs-Ag)
* Normal or elevated ALT/GTP values at screening
* At known diabetes mellitus or hypertension an ophthalmologic examination must be performed
* Liver biopsy within the last 12 months must confirm the diagnoses of a chronic hepatitis
* A confirmation must be given that sexually active patients practice a save method of contraception during the therapy and 6 (women) to 7 (men) months after the therapy

Exclusion Criteria:

* Age < 18 years, > 70 years
* Previous treatment of hepatitis c with (Peg)Interferon alfa or (Peg)Interferon alfa/Ribavirin
* Patients with organ transplantations other than cornea or hair
* Infection with HCV genotype 2,3,4,5 or 6
* Pregnant or nursing women
* Any other reason for the liver disease than chronic hepatitis C
* Suspected hypersensitivity to Interferon, Peginterferon or Ribavirin
* Participation in a clinical trial or treatment with an investigational product 30 days before inclusion in this study
* Patients with any kind of hemoglobinopathy
* Documented liver disease in advanced state Liver cirrhosis Child B and C
* Each known and existing clinical conditions that might challenge the participation or completion of this clinical trial as depressions, psychosis, severe psychiatric diseases, suicide ideations CNS traumata or cramps which need medicamentous treatment
* Relevant cardiovascular dysfunctions in the last 6 months or patients with clinically relevant changes in the ECG
* Insufficiently adjusted diabetes mellitus
* Severe chronic lung diseases (as e.g. COPD)
* Immunologic diseases or autoimmune-diseases or any other disease which demand a longtime treatment with corticosteroids during this clinical trial
* Clinically relevant gout
* Abuse of drugs, alcohol or pharmaceuticals
* Patient with clinically relevant changes of the retina
* Missing ability or willingness to understand the purpose of this study or to give a written consent for participating in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2006-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Sustained viral response (HCV RNA negativity 24 weeks after end of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Sarrazin, MD, PhD, Study Chair — University Hospital, Saarland
Locations (22):
- Germany (22):
  - Medizinische Universitätsklinik Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinik Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Uniklinikum Erlangen, Erlangen, Bavaria
  - Klinikum Großhadern, München, Bavaria
  - Technische Universität München, München, Bavaria
  - Klinikum der Universität Würzburg, Würzburg, Bavaria
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg, Hamburg
  - Klinikum der J.W.-Goethe-Universität, Frankfurt am Main, Hesse
  - Praxis für Innere Medizin, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitätsklinikum Aachen, Aachen, Nordrhein.Westfalen
  - St. Josef-Hospital, Bochum, North Rhine-Westphalia
  - Universität zu Köln, Cologne, North Rhine-Westphalia
  - Gemeinschaftspraxis, Düsseldorf, North Rhine-Westphalia
  - Medizinische Universitäts-Klinik Essen, Essen, North Rhine-Westphalia
  - Universitätsklinikum der J. Gutenberg Universität, Mainz, Rhineland-Palatinate
  - Universitätsklinikum des Saarlandes, Homburg / Saar, Saarland
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Christian-Albrechts-Universität zu Kiel, Kiel, Schleswig-Holstein
  - Hepatologische Schwerpunktpraxis, Berlin, State of Berlin
  - Charité, Campus Virchow-Klinikum, Berlin, State of Berlin

REFERENCES:
- [Derived] Sarrazin C, Schwendy S, Moller B, Dikopoulos N, Buggisch P, Encke J, Teuber G, Goeser T, Thimme R, Klinker H, Boecher WO, Schulte-Frohlinde E, Prinzing R, Herrmann E, Zeuzem S, Berg T. Improved responses to pegylated interferon alfa-2b and ribavirin by individualizing treatment for 24-72 weeks. Gastroenterology. 2011 Nov;141(5):1656-64. doi: 10.1053/j.gastro.2011.07.019. Epub 2011 Jul 22. PMID 21784046